CLINICAL TRIAL: NCT07096271
Title: Better Together: A Relationship Enrichment Program Targeting Transdiagnostic Interpersonal Emotion Regulation Among Military Couples
Brief Title: Get Better Together: Relationship Education For Military Couples
Acronym: GBT RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USUHS.2022-100; HT94252410843 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Emotion Regulation; Relationship Conflict; Suicide Risk; Alcohol Use; Intimate Partner Violence (IPV); Relationship Distress; Interpersonal Emotion Regulation
Keywords: Behavioral: Get Better Together (GBT); military; intimate relationships; suicide prevention; primary prevention; emotion regulation; relationship education; interpersonal emotion regulation
MeSH Terms: conditions — Emotional Regulation; Alcohol Drinking; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Get Better Together (GBT) (Experimental): Participants assigned to this arm will attend an in-person weekend retreat where they receive approximately 10 hours of structured curriculum focused on equipping couples with evidence informed strategies to cope with stress as a team, improve emotion regulation, and reduce conflict.
  GBT includes modules on emotion awareness, acceptance, reappraisal, constructive problem solving, and communication. The format integrates didactic material, videos, group discussions, and couples' skill practice. All materials and delivery methods have been tailored for military populations based on extensive stakeholder input and field testing.
  Interventions: Behavioral: Get Better Together (GBT)
- Control Group (No Intervention): Couples in the control group will not receive any structured relationship enrichment programming (e.g., retreats or workshops) during the 6-month follow-up period. After the 6-month follow-up period, couples in the control group will be provided access to ePREP, a self-paced on line version of the PREP curriculum.

INTERVENTIONS:
Behavioral: Get Better Together (GBT) — Get Better Together is a couple-based, primary prevention program designed to reduce risk for suicidal thoughts and behaviors, problematic alcohol use, and intimate partner violence by addressing two transdiagnostic drivers: emotion dysregulation and relationship conflict. The intervention is an adaptation of the empirically supported Prevention and Relationship Enhancement Program (PREP), modified in collaboration with military stakeholders to meet the unique cultural and contextual needs of military couples.
  The GBT curriculum includes approximately 10 hours of structured content presented using didactic instruction, video demonstrations, group discussions, and guided couple exercises. Skills focus on interpersonal emotion regulation (e.g., emotion identification, acceptance, reappraisal, and problem solving) and evidence-based communication strategies (e.g., structured communication strategies, conflict de-escalation).
  Arms: Get Better Together (GBT)

SUMMARY:
This study is testing a program called Get Better Together, a relationship education program designed to help military couples effectively navigate life stressors as a team. The goal is to find out if attending Get Better Together improves mental health and relationship skills, and reduces problems like alcohol misuse, aggression, and suicide risk. Couples who join the study will be randomly placed into one of two groups. One group will attend Get Better Together at a weekend retreat. The other group will continue their usual activities and later receive access to an online relationship education program. All participants will complete surveys before the retreat and again 2, 4, and 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Couple is in a committed romantic relationship of at least six months
* At least one partner is a military Service member on active duty
* Both partners are age 18 or older
* Couple has not previously attended a relationship enrichment retreat or workshop together (e.g., CREDO, Strong Bonds, BSRT). This does not include couples therapy or pre-marital counseling.

Exclusion Criteria:

* One or both partners decline to provide informed consent
* Required command endorsement for retreat attendance is not received (for Service members E-6 and below)
* Couple is unable or unwilling to attend any of the scheduled retreats during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Suicide Cognitions | Baseline, 2-month, 4-month, and 6-month follow-up
  Assessed using the Suicide Cognition Scale-Revised (SCS-R), a 16-item validated self-report measure capturing cognitive risk factors for suicidal behavior. Scores range from 0 to 64, with higher scores reflect greater risk.
Alcohol Misuse | Baseline, 2-month, 4-month, and 6-month follow-up
  Measured using the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C), a 3-item measure designed to identify hazardous drinking. Scores range from 0 to 12, with higher scores reflect greater likelihood of drinking affecting one's health and safety.
Intimate Partner Violence | Baseline, 2-month, 4-month, and 6-month follow-up
  Measured using the Revised Conflict Tactics Scale-Short Form (CTS2S), a 20-item measure assessing multiple types of relationship abuse. Dichotomous scores will indicate the presence of any form of abuse. Dichotomous subscale scores will indicate the presence of assault, injury, psychological aggression, or sexual coercion.

SECONDARY OUTCOMES:
Emotion Dysregulation | Baseline, 2-month, 4-month, and 6-month follow-up
  Measured using the Difficulties in Emotion Regulation Scale - 18 Item (DERS-18), which assesses six dimensions of emotion dysregulation: awareness, clarity, nonacceptance, impulse, goals, and strategies. Total scores range from 18 to 90, with higher scores indicating more severe difficulties regulating one's emotions.
Relationship Conflict | Baseline, 2-month, 4-month, and 6-month follow-up
  Evaluated using the Ineffective Arguing Inventory (IAI), an 8-item scale measuring perceived patterns of unresolved conflict and communication breakdown in romantic relationships. Total scores range from 8 to 40, with higher scores indicating a higher degree of ineffective communication.
Interpersonal Emotion Regulation with Romantic Partner | Baseline, 2-month, 4-month, and 6-month follow-up
  Measured using the Dyadic Coping Inventory (DCI), an 37-item self-report measure assessing how couples communicate stress and cope together (supportive, delegated, negative, and joint coping). Total scores range from 37 to 185, with higher scores indicated higher levels of dyadic coping.
Relationship Functioning | Baseline, 2-month, 4-month, and 6-month follow-up
  Assessed using the Revised Dyadic Adjustment Scale (RDAS), a 14-item self-report measure evaluating relationship functioning across three domains: Dyadic Consensus, Dyadic Satisfaction, and Dyadic Cohesion. Items assess agreement on relationship issues, frequency of shared activities, and satisfaction with the relationship. Total scores range from 0 to 69, with higher scores indicating greater relationship satisfaction.

OTHER OUTCOMES:
Military Readiness (active-duty participants only) | Baseline, 2-month, 4-month, and 6-month follow-up
  Measured using items adapted from the 2017 Workplace and Equal Opportunity Survey of Active Duty Members (Office of People Analytics, 2018), a DoD standardized survey tool. Items assess key indicators of readiness, including self intent to remain in the military. Items use Likert-type scales appropriate to each domain (e.g., "Very poorly prepared" to "Very well prepared"). The items are designed to be used independently rather than as a single composite scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Carter, Ph.D., Principal Investigator — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected through self-report surveys will be shared, including composite scores, coded record based variables (e.g., derived from DoD administrative or health records), and contextual data related to study implementation. No shared data will include personally identifiable information (PII) or protected health information (PHI). All data sharing will comply with IRB, institutional, and federal requirements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 12 months after publication of primary outcomes. No planned end date.
Access Criteria: Access to de-identified trial data may be provided to qualified researchers. Requests are subject to review and require a brief proposal and a signed Data Use Agreement outlining appropriate safeguards and data handling procedures.

DOCUMENTS (1):
  • Informed Consent Form (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT07096271/ICF_000.pdf